CLINICAL TRIAL: NCT00138762
Title: A Phase 3, Double Blind, Placebo-Controlled, Randomized, Parallel Group, Multicenter Study of the Efficacy, Safety and Tolerability of Fixed Combination Torcetrapib/Atorvastatin Administered Orally Once Daily for 6 Months, Compared to Atorvastatin Alone or Placebo in Subjects With Mixed Dyslipidemia (Fredrickson Types IIa and IIb).
Brief Title: A Study of Torcetrapib/Atorvastatin vs Atorvastatin Alone or Placebo in Patients With High Cholesterol
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5091018
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias | interventions — torcetrapib; Atorvastatin

INTERVENTIONS:
Drug: torcetrapib/atorvastatin
Drug: atorvastatin
Drug: placebo

SUMMARY:
The Torcetrapib project was terminated on December 2, 2006 due to safety findings.

A study to look at lipid levels in subjects taking the study drug, Atorvastatin alone or placebo.

DETAILED DESCRIPTION:
For additional information please call: 1-800-718-1021

ELIGIBILITY:
Inclusion Criteria:

* subjects with elevated cholesterol

Exclusion Criteria:

* Women who are pregnant or lactating, or planning to become pregnant.
* Intolerance to statin therapy resulting in withdrawal
* Subjects taking any drugs known to be associated with an increased risk of myositis in combination with HMG-CoA reductase inhibitors
* Subjects with any other medical condition or laboratory abnormality which could affect subject safety, preclude evaluation of response, or render unlikely that the subject would complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3800
Dates: Start 2004-07; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
LDL and HDL levels

SECONDARY OUTCOMES:
other lipid parameters

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (154):
- United States (96):
  - Pfizer Investigational Site, Mobile, Alabama
  - Pfizer Investigational Site, Mesa, Arizona
  - Pfizer Investigational Site, Oro Valley, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Sun City, Arizona
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, Carmichael, California
  - Pfizer Investigational Site, Concord, California
  - Pfizer Investigational Site, Greenbrae, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Mission Viejo, California
  - Pfizer Investigational Site, Sacramento, California
  - Pfizer Investigational Site, Santa Ana, California
  - Pfizer Investigational Site, Stockton, California
  - Pfizer Investigational Site, Thouasand Oaks, California
  - Pfizer Investigational Site, Tustin, California
  - Pfizer Investigational Site, Upland, California
  - Pfizer Investigational Site, Walnut Creek, California
  - Pfizer Investigational Site, Westlake Village, California
  - Pfizer Investigational Site, Boulder, Colorado
  - Pfizer Investigational Site, Waterbury, Connecticut
  - Pfizer Investigational Site, Newark, Delaware
  - Pfizer Investigational Site, Coral Gables, Florida
  - Pfizer Investigational Site, Ft. Pierce, Florida
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Jupiter, Florida
  - Pfizer Investigational Site, Lake Worth, Florida
  - Pfizer Investigational Site, Melbourne, Florida
  - Pfizer Investigational Site, Palm Bay, Florida
  - Pfizer Investigational Site, Sebastian, Florida
  - Pfizer Investigational Site, Stuart, Florida
  - Pfizer Investigational Site, Vero Beach, Florida
  - Pfizer Investigational Site, Wellington, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Creve Coevr, Illinois
  - Pfizer Investigational Site, Peoria, Illinois
  - Pfizer Investigational Site, Rockford, Illinois
  - Pfizer Investigational Site, Iowa City, Iowa
  - Pfizer Investigational Site, Kansas City, Kansas
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Erlanger, Kentucky
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Covington, Louisiana
  - Pfizer Investigational Site, Slidell, Louisiana
  - Pfizer Investigational Site, Scarborough, Maine
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Bethesda, Maryland
  - Pfizer Investigational Site, Elkton, Maryland
  - Pfizer Investigational Site, Jackson, Mississippi
  - Pfizer Investigational Site, Jefferson City, Missouri
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, Billings, Montana
  - Pfizer Investigational Site, Lincoln, Nebraska
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Endwell, New York
  - Pfizer Investigational Site, Lake Success, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Williamsville, New York
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Concord, North Carolina
  - Pfizer Investigational Site, Fayetteville, North Carolina
  - Pfizer Investigational Site, Monroe, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Elyria, Ohio
  - Pfizer Investigational Site, Olmsted, Ohio
  - Pfizer Investigational Site, Westlake, Ohio
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Beaverton, Oregon
  - Pfizer Investigational Site, Hillsboro, Oregon
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Warwick, Rhode Island
  - Pfizer Investigational Site, Greer, South Carolina
  - Pfizer Investigational Site, Spartanburg, South Carolina
  - Pfizer Investigational Site, Kingsport, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Beaumont, Texas
  - Pfizer Investigational Site, Bryan, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, The Colony, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Newport News, Virginia
  - Pfizer Investigational Site, Norfolk, Virginia
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Renton, Washington
  - Pfizer Investigational Site, Yakima, Washington
  - Pfizer Investigational Site, Milwaukee, Wisconsin
  - Pfizer Investigational Site, Oregon, Wisconsin
- Belgium (8):
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Dottignies
  - Pfizer Investigational Site, Ham
  - Pfizer Investigational Site, Hasselt
  - Pfizer Investigational Site, Hoeilaart
  - Pfizer Investigational Site, La Louvière
  - Pfizer Investigational Site, Leuven
  - Pfizer Investigational Site, Wilsele
- Germany (15):
  - Pfizer Investigational Site, Beckum
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Bochum
  - Pfizer Investigational Site, Erlangen
  - Pfizer Investigational Site, Essen
  - Pfizer Investigational Site, Feldafing
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Heidelberg
  - Pfizer Investigational Site, Homburg/Saar
  - Pfizer Investigational Site, Karlsruhe
  - Pfizer Investigational Site, Künzing
  - Pfizer Investigational Site, Nuremberg
  - Pfizer Investigational Site, Offenbach
  - Pfizer Investigational Site, Rodgau
  - Pfizer Investigational Site, Schwerin
- Mexico (5):
  - Pfizer Investigational Site, México, D.f.
  - Pfizer Investigational Site, Tlalpan, D.f.
  - Pfizer Investigational Site, Mexico City, Mexico City
  - Pfizer Investigational Site, Monterrey, Nuevo León
  - Pfizer Investigational Site, Puebla City, Puebla
- Norway (13):
  - Pfizer Investigational Site, Bekkestua
  - Pfizer Investigational Site, Elverum
  - Pfizer Investigational Site, Hønefoss
  - Pfizer Investigational Site, Jessheim
  - Pfizer Investigational Site, Kongsberg
  - Pfizer Investigational Site, Lena
  - Pfizer Investigational Site, Lierskogen
  - Pfizer Investigational Site, Molde
  - Pfizer Investigational Site, Moss
  - Pfizer Investigational Site, Oslo
  - Pfizer Investigational Site, Roverud
  - Pfizer Investigational Site, Skedsmokorset
  - Pfizer Investigational Site, Tromsø
- South Korea (2):
  - Pfizer Investigational Site, Seoul
  - Pfizer Investigational Site, Suwon
- Sweden (6):
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Jarfalla
  - Pfizer Investigational Site, Linköping
  - Pfizer Investigational Site, Örebro
  - Pfizer Investigational Site, Strängnäs
  - Pfizer Investigational Site, Umeå
- United Kingdom (9):
  - Pfizer Investigational Site, Penzance, Cornwall
  - Pfizer Investigational Site, Woolwell, Plymouth, Devon
  - Pfizer Investigational Site, Middlesex, Harrow
  - Pfizer Investigational Site, Garston, Hertfordshire
  - Pfizer Investigational Site, Blackpool, Lancashire
  - Pfizer Investigational Site, Blackpool, Lancs. Fy3 7dq
  - Pfizer Investigational Site, Addlestone, Surrey
  - Pfizer Investigational Site, East Horsley, Leatherhead, Surrey
  - Pfizer Investigational Site, Warminster, Wiltshire